CLINICAL TRIAL: NCT01702974
Title: Immune Reconstitution in HIV Disease Using Antimicrobial Treatment With Vitamin D and Phenylbutyrate
Brief Title: Immune Reconstitution in HIV Disease (IREHIV)
Acronym: IREHIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Addis Ababa University (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Susanna Brighenti, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IREHIV-2012
Record Dates: First submitted 2012-09-25; First posted 2012-10-10 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV; cholecalciferol; sodium phenylbutyrate; antimicrobial peptides; immune response; inflammation
MeSH Terms: conditions — HIV Infections; Inflammation | interventions — Vitamin D; Cholecalciferol; 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate) (Active Comparator): Dose of interventions: 5,000 IU of vitamin D (cholecalciferol tablets) once daily and 500 mg PBA (sodium phenylbutyrate tablets) twice daily for 16 weeks.
  Interventions: Drug: vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate)
- Placebo tablets (Placebo Comparator): Placebo tablets for vitamin D once daily and placebo tablets for PBA (phenylbutyrate) twice daily for 16 weeks.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate) — Dose of interventions: 5,000 IU of vitamin D (cholecalciferol tablets) once daily and 500 mg PBA (sodium phenylbutyrate tablets) twice daily for 16 weeks.
  Arms: Vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate)
Drug: Placebo tablets — Placebo tablets for vitamin D once daily and placebo tablets for PBA (phenylbutyrate) twice daily for 16 weeks.
  Arms: Placebo tablets

SUMMARY:
The aim with this study is to provide immunotherapy with vitamin D and phenylbutyrate to treatment-naive HIV infected patients to induce important antimicrobial defence mechanisms and decreased inflammation.

ELIGIBILITY:
Inclusion Criteria:

Adult patients >18 years not subjected to HAART.

HIV-1 infected patients with CD4 T cells counts >200 cells/ml.

Detectable plasma viral loads >1000 copies/ml.

Exclusion Criteria:

Patients on HAART or other antimicrobial drugs (including bactrim).

Antimicrobial drug treatment in the past month.

Patients with medical contra-indication for biopsy such as bleeding tendencies.

Hypercalcaemia (serum calcium > 3,0 mmol/L) identified at baseline.

Pregnant and breast feeding women.

Any known liver or kidney function abnormality, malignancy or patients treated with cardiac glycosides.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
HIV viral load | 0 (baseline) compared to 16 weeks.
  Plasma HIV viral load will be used to monitor efficacy of vitamin D and phenylbutyrate treatment among treatment-naïve HIV patients at the time of diagnosis (time point 0) and at 4, 8, 16 and 24 weeks after initiation of antimicrobial treatment with vitamin D and phenylbutyrate. The primary endpoint will be assessed at 16 weeks compared to baseline (time point 0).

SECONDARY OUTCOMES:
Clinical secondary endpoints | 0, 4, 8, 16, 24 weeks.
  Overall clinical symptoms.
  Body mass index (BMI).
  Mid upper arm circumference (MUAC).
Laboratory secondary endpoints | 0, 4, 8, 16, 24 weeks.
  HIV viral load (0, 4, 8, 24 weeks).
  Peripheral CD4/CD8 T cell counts.
  Plasma levels of vitamin D, LL-37, sCD14, LPS, 16S RNA and cytokine/chemokine profiles.
  Calprotectin in feces.
  Inflammation and microbial translocation in colon punch biopsies (0 and 16 weeks).
  Functional studies of immune cells (PBMCs).

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Brighenti, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Black Lion Hospital (BLH), Addis Ababa University, Faculty of Medicine, Addis Ababa, Lideta Sub City, Ethiopia

REFERENCES:
- [Derived] Missailidis C, Sorensen N, Ashenafi S, Amogne W, Kassa E, Bekele A, Getachew M, Gebreselassie N, Aseffa A, Aderaye G, Andersson J, Brighenti S, Bergman P. Vitamin D and Phenylbutyrate Supplementation Does Not Modulate Gut Derived Immune Activation in HIV-1. Nutrients. 2019 Jul 21;11(7):1675. doi: 10.3390/nu11071675. PMID 31330899
- [Derived] Ashenafi S, Amogne W, Kassa E, Gebreselassie N, Bekele A, Aseffa G, Getachew M, Aseffa A, Worku A, Hammar U, Bergman P, Aderaye G, Andersson J, Brighenti S. Daily Nutritional Supplementation with Vitamin D(3) and Phenylbutyrate to Treatment-Naive HIV Patients Tested in a Randomized Placebo-Controlled Trial. Nutrients. 2019 Jan 10;11(1):133. doi: 10.3390/nu11010133. PMID 30634590